CLINICAL TRIAL: NCT03303599
Title: Real World Evidence of the Effectiveness and Clinical Practice Use of Glecaprevir Plus Pibrentasvir in Patients With Chronic Hepatitis C Genotypes 1 to 6
Brief Title: Study of the Effectiveness and Clinical Practice Use of Glecaprevir Plus Pibrentasvir in Patients With Chronic Hepatitis C Genotypes 1 to 6
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P17-094
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C; Sustained Virological Response; Chronic Hepatitis C genotype 1; Chronic Hepatitis C genotype 2; Chronic Hepatitis C genotype 3; Chronic Hepatitis C genotype 4; Chronic Hepatitis C genotype 5; Chronic Hepatitis C genotype 6
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCV Genotypes 1, 2, 3, 4, 5, or 6 participants: Participants receiving combination therapy with the glecaprevir plus pibrentasvir (GLE/PIB) regimen according to standard of care, international guidelines and in line with the current local label.

SUMMARY:
The interferon- and ribavirin- (RBV) free combination regimen of glecaprevir plus pibrentasvir (GLE/PIB) for the treatment of genotypes 1 to 6 of chronic hepatitis C (CHC) viral infection has been shown to be safe and effective in randomized controlled clinical trials.

This observational study is an effectiveness research examining the regimen of GLE/PIB, used according to local label, under real world conditions in a clinical practice patient population.

ELIGIBILITY:
Inclusion Criteria:

* Participants are treatment-naïve or treatment-experienced with pegylatedinterferon (pegIFN), or IFN, and/or ribavirin (RBV) and/or sofosbuvir (PRS) with confirmed chronic hepatitis C (CHC), genotypes 1, 2, 3, 4, 5, or 6, with or without compensated cirrhosis, receiving combination therapy with the all oral glecaprevir plus pibrentasvir (GLE/PIB) regimen according to standard of care, international guidelines and in line with the current local label.
* Participants may be enrolled up to 4 weeks after treatment initiation
* Participants must not be participating or intending to participate in a concurrent interventional therapeutic trial.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving GLE/PIB who have started the treatment combination recommended in the current local label for their disease characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 2118 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving sustained virological response 12 weeks post-treatment (SVR12) | 12 weeks (i.e. at least 70 days) after the last dose of Glecaprevir plus Pibrentasvir
  SVR12 defined as the hepatitis C virus (HCV) ribonucleic acid (RNA) level less than the lower limit of quantification 12 weeks after the last dose of Glecaprevir plus Pibrentasvir

SECONDARY OUTCOMES:
Percentage of Participants Taking Concomitant Medications | Up to approximately 28 weeks
  The percentage of participants taking concomitant medications from the decision to initiate treatment through 12 weeks after the last dose of glecaprevir plus pibrentasvir.
Percentage of Glecaprevir plus Pibrentasvir (GLE/PIB) Doses Taken out of that Prescribed | Up to approximately 16 weeks
  The percentage of GLE/PIB doses taken by participant in relation to the prescribed target dose (number of pills taken out of the number of pills that should have been taken).
Changes from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Up to 16 weeks
  Among participants with renal impairment, changes from baseline during treatment in estimated glomerular filtration rate (eGFR determined by Modification of Diet in Renal Disease [MDRD] equation).
Number of Healthcare Resource Utilization (HCRU) | Up to approximately 28 weeks
  Health Care Resource Utilization (HCRU) for a participant will be the total number of visits/touchpoints (face to face or phone call) with an Health Care Provider (HCP) or designee in relation to their HCV infection during the study.
Percentage of Participants Using Each Treatment Regimen | Up to 16 weeks
  Percentage of participants using each treatment regimen (intended treatment duration of 8, 12, or 16 weeks)
Percentage of Participants with Co-morbidities | Baseline (Day 1)
  The percentage of participants with co-morbidities at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (156):
- Austria (8):
  - Klinikum Klagenfurt am Woerthersee, Apotheke /ID# 169931, Klagenfurt, Carinthia
  - University Hospital St. Polten /ID# 169918, Sankt Pölten, Lower Austria
  - Medizinische Universität Graz /ID# 169932, Graz, Styria
  - Landeskrankenhaus Hall /ID# 169930, Hall in Tirol, Tyrol
  - KH der Elisabethinen Linz GmbH /ID# 169915, Linz, Upper Austria
  - Landeskrankenhaus /ID# 169922, Innsbruck
  - Wilhelminenspital der Stadt Wien /ID# 169914, Vienna
  - Klinikum Wels - Grieskirchen /ID# 169916, Wels
- Belgium (19):
  - Uza /Id# 170960, Edegem, Antwerpen
  - UCL Saint-Luc /ID# 170964, Woluwe-Saint-Lambert, Brussels Capital
  - Algemeen Stedelijk Ziekenhuis /ID# 170876, Aalst, Oost-Vlaanderen
  - UZ Gent /ID# 170922, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 170921, Leuven, Vlaams-Brabant
  - Centre Hospitalier de Wallonie Picarde /ID# 200822, Tournai, Wallonne, Region
  - Zna /Id# 170927, Antwerp
  - CHU Saint-Pierre /ID# 170920, Brussels
  - CHU Brugmann /ID# 170956, Brussels
  - Hopital Erasme /ID# 170918, Brussels
  - Z.O.L - Campus St. Jan /ID# 171058, Genk
  - AZ Middelares Gent /ID# 170874, Ghent
  - Jessa Ziekenhuis /ID# 170958, Hasselt
  - AZ Groeninge /ID# 170931, Kortrijk
  - Centre Hospitalier Universitaire du Sart Tilman CHU de Liege /ID# 170930, Liège
  - CHC Liege /ID# 170926, Liège
  - CHU Ambroise Pare /ID# 171107, Mons
  - Clinique Edith Cavell /ID# 170932, Uccle
  - CHU Dinant Godinne /ID# 170929, Yvoir
- France (49):
  - CHR Orleans - Hopital de la Source /ID# 202360, Orléans, Centre-Val de Loire
  - CH Georges Renon /ID# 202737, Niort, Deux-Sevres
  - CHU de Besancon - Jean Minjoz /ID# 208502, Besançon, Doubs
  - CHU Dupuytren /ID# 202514, Limoges, Franche-Comte
  - Hopital Haut-Lévêque /ID# 202501, Pessac, Gironde
  - Hopital Purpan /ID# 202357, Toulouse, Haute-Garonne
  - Hopital Purpan /ID# 204201, Toulouse, Haute-Garonne
  - CH Annecy Genevois Site Annecy /ID# 202804, Epagny Metz Tessy, Haute-Savoie
  - CH Spécialisé Esquirol /ID# 204522, Limoges, Haute-Vienne
  - Centre Hospitalier de Béziers /ID# 202948, Béziers, Herault
  - Hopital Saint Eloi /ID# 202512, Montpellier, Herault
  - Hopital Broussais /ID# 202677, St-Malo, Ille-et-Vilaine
  - CHU NANCY - Hopital Brabois Adultes /ID# 202570, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hopital de la Timone /ID# 202792, Marseille, Provence-Alpes-Côte d'Azur Region
  - Charles Nicolle CHU Rouen /ID# 203518, Rouen, Seine-Maritime
  - Centre Hosp Intercommunal de Creteil /ID# 202566, Créteil, Val-de-Marne
  - Cabinet medical /ID# 202794, Aix-en-Provence
  - CHU d'Angers /ID# 202500, Angers
  - Clinique du Tondu /ID# 207508, Bordeaux
  - Centre Endo Nord Isere /ID# 204181, Bourgoin
  - Hopital de la Cavale Blanche /ID# 202640, Brest
  - Hopital Antoine Beclere /ID# 202676, Clamart
  - CHU Estaing /ID# 202949, Clermont-Ferrand
  - Hopital Henri Mondor /ID# 202806, Créteil
  - Centre Hospitalier Universitaire de Grenoble - Hopital Michallon /ID# 202957, Grenoble
  - CH d'Hyeres /ID# 202515, Hyères
  - Dr. Cuissard, Le Port, FR /ID# 203487, Le Port
  - C.H. de Bretagne Sud /ID# 202362, Lorient
  - Hopital de la Croix Rousse /ID# 203071, Lyon
  - Hopital Edouard Herriot /ID# 203149, Lyon
  - Hopital Europeen /ID# 205073, Marseille
  - Hopital Saint Joseph /ID# 202519, Marseille
  - Cabinet Medical, Boyer Darrigr /ID# 202050, Nanterre
  - Hopital l'Archet 2 /ID# 205295, Nice
  - CHU Nimes /ID# 208200, Nîmes
  - Hopital Bichat-Claude Bernard /ID# 202513, Paris
  - Hopital Saint Antoine /ID# 202565, Paris
  - Hopital Pitie Salpetriere /ID# 202364, Paris
  - Centre Hospitalier PERPIGNAN /ID# 205762, Perpignan
  - Hopital Robert Debre /ID# 202953, Reims
  - Gastrodoc /Id# 206290, Saint-Jean-de-Védas
  - Institut Arnault Tzanck /ID# 202363, Saint-Laurent-du-Var
  - Cabinet Medical, Dr. Constant, /ID# 202361, Toulon
  - Clinique Amroise Pare /ID# 205064, Toulouse
  - Hopital Joseph Ducuing /ID# 205666, Toulouse
  - Ctre Hospitalier de Tourcoing /ID# 202358, Tourcoing
  - Ctre Hospitalier de Tourcoing /ID# 202805, Tourcoing
  - Hopital Paul Brousse /ID# 202623, Villejuif
  - Hopital Beaujon /ID# 202675, Clichy, Île-de-France Region
- Greece (10):
  - General Hospital of Athens Laiko /ID# 206421, Athens, Attica
  - General Oncological Hospital of Kifisia Oi Agioi Anargyroi /ID# 206419, Kifissia, Attica
  - Tzaneio general hospital of Piraeus /ID# 208828, Piraeus, Attica
  - Papageorgiou General Hospital Thessaloniki /ID# 207980, Nea Efkarpia, Thessaloniki
  - Gen Univ Hosp Alexandroupolis /ID# 206416, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 206414, Athens
  - General Hospital Nikaias-Piraeus St. Panteleimon /ID# 206420, Pireaus
  - Bioclinic Thessaloniki /ID# 207981, Thessaloniki
  - University Gen Hosp AHEPA /ID# 209961, Thessaloniki
  - Interbalkan Medical Center /ID# 206417, Thessaloniki
- Israel (15):
  - Soroka Medical Center /ID# 169321, Beersheba, Southern District
  - HaEmek Medical Center /ID# 169318, Afula
  - Assaf Harofeh Medical Center /ID# 169370, Be’er Ya‘aqov
  - Maccabi Health Services /ID# 169372, GUSH DAN
  - Hillel Yaffe Medical Center /ID# 169368, Hadera
  - Rambam Medical Center /ID# 169316, Haifa
  - Bnai Zion Medical Center /ID# 169358, Haifa
  - Carmel Medical Center /ID# 169309, Haifa
  - Shaare Zedek Medical Center /ID# 169329, Jerusalem
  - Gastroenterology Institute, Division of Medicine /ID# 169360, Jerusalem
  - Meir Medical Center /ID# 169327, Kfar Saba
  - Galilee Medical Center /ID# 169325, Nahariya
  - Rabin Medical Center /ID# 169320, Petah Tikva
  - Sheba Medical Center /ID# 169365, Ramat Gan
  - Tel Aviv Medical Center /ID# 169313, Tel Aviv
- Italy (29):
  - AOU Federico II /ID# 168131, Naples, Campania
  - Ospedale Sant Orsola Malpighi /ID# 168127, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Policlinico di Modena /ID# 168711, Modena, Emilia-Romagna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 168137, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 168138, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 168712, Milan, Lombardy
  - IBD Center - IRCCS Istituto Clinico Humanitas /ID# 169353, Rozzano, Milano
  - AOU Citta della Salute Scienza /ID# 168142, Turin, Piedmont
  - Fondazione PTV Policlinico Tor Vergata /ID# 168709, Rome, Roma
  - Università Cattolica Sacro Cuore /ID# 168781, Rome, Roma
  - Policlinico Paolo Giaccone /Id# 168134, Palermo, Sicily
  - Azienda Universitaria Ospedali /ID# 168129, Bari
  - AOU di Cagliari - Presidio di /ID# 168132, Cagliari
  - A.O.U Sant'Anna di Ferrara /ID# 168714, Ferrara
  - AOU Riuniti di Foggia /ID# 168143, Foggia
  - Ospedale SM Goretti /ID# 169257, Latina
  - A.O.U. Policlinico G. Martino /ID# 168139, Messina
  - Ospedale S. Carlo Borromeo /ID# 168144, Milan
  - Azienda Ospedaliera Luigi Sacc /ID# 168136, Milan
  - Azienda Ospedaliera Luigi Sacc /ID# 168140, Milan
  - Azienda Ospedaliera di Rilievo /ID# 168141, Naples
  - AO Domenico Cutugno /ID# 168133, Napoli
  - Universita degli Studi della /ID# 168135, Napoli
  - Azienda Ospedaliera Maggiore d /ID# 168710, Novara
  - Azienda Ospedaliera di Padova /ID# 168125, Padua
  - Azienda Ospedaliera di Padova /ID# 168126, Padua
  - Azienda Ospedaliero - Universi /ID# 168130, Pisa
  - IRCCS Lazzaro Spallanzani /ID# 169234, Rome
  - AOU OO. RR. San Giovanni di Di /ID# 168715, Salerno
- Poland (14):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II /ID# 208451, Krakow, Lesser Poland Voivodeship
  - Specjalistyczny Szpital im. dra Alfreda Sokolowskiego /ID# 208862, Wałbrzych, Lower Silesian Voivodeship
  - NZOZ - Lubuska Specjalistyczna Poradnia Chorób Wątroby Sp. z o.o. /ID# 208449, Zielona GORA, Lower Silesian Voivodeship
  - Szpital Wojewodzki w Opolu /ID# 208444, Opole, Opole Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku /ID# 208604, Bialystok, Podlaskie Voivodeship
  - Szpital Specjalistyczny W Chorzowie /Id# 209129, Chorzów, Silesian Voivodeship
  - NZOZ All-Medicus /ID# 208452, Katowice, Silesian Voivodeship
  - ID Clinic /ID# 208332, Mysłowice, Silesian Voivodeship
  - Wojewodzki Szpital Obserwacyjn /ID# 209345, Bydgoszcz
  - Wojewódzki Szpital Zespolony w Kielcach /ID# 210569, Kielce
  - Wojewodzki Szpit Bieganskiego /ID# 208445, Lodz
  - Wojewodzki Szpit Bieganskiego /ID# 209608, Lodz
  - MED-FIX Centrum Medyczne Sp. z /ID# 208453, Warsaw
  - NZOZ Przychodnia Specjalistycz /ID# 208334, Żychlin, Łódź Voivodeship
- Portugal (6):
  - Centro Hospitalar Barreiro Montijo, EPE /ID# 211267, Barreiro, Lisbon District
  - Centro Hospitalar Vila Nova Gaia/Espinho, EPE /ID# 208195, Vila Nova de Gaia, Porto District
  - Hospital Garcia de Orta, E.P.E /ID# 207717, Almada, Setúbal District
  - Centro Hospitalar Universitário Lisboa Central, EPE - Hospital Curry Cabral /ID# 208463, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 207910, Lisbon
  - Centro Hospitalar do Porto EPE /ID# 207733, Porto
- Switzerland (6):
  - Hopitaux Universitaires de Geneve /ID# 203435, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen /ID# 201025, Sankt Gallen, Canton of St. Gallen
  - Inselspital, Universitaetsklinik /ID# 201022, Bern
  - Fondazione Epatocentro Ticino /ID# 201024, Lugano
  - Hopital Neuchatelois /ID# 201026, Neuchâtel
  - Universitaetsspital Zuerich /ID# 201023, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vera J, Gomes A, Povoas D, Seixas D, Maltez F, Pedroto I, Maia L, Mota M, Vieira MJ, Manata MJ, Ferreira P, Lino S, Pereira Guedes T, Barradas V, Marques N. Real-World Effectiveness and Safety of Glecaprevir/Pibrentasvir for the Treatment of Chronic Hepatitis C: A Prospective Cohort Study in Portugal. Acta Med Port. 2024 May 2;37(5):323-333. doi: 10.20344/amp.19178. Epub 2024 Feb 7. PMID 38325411
- [Derived] Aghemo A, Horsmans Y, Bourgeois S, Bondin M, Gschwantler M, Hofer H, Semmo N, Negro F, Zhang Z, Marcinak J, Veitsman E, Hazzan R, Mimidis K, Goulis I, Marques N, Flisiak R, Mazur W, Roncero C, Marra F, Pageaux GP, Asselah T, Lampertico P. Real-World Outcomes in Historically Underserved Patients with Chronic Hepatitis C Infection Treated with Glecaprevir/Pibrentasvir. Infect Dis Ther. 2021 Dec;10(4):2203-2222. doi: 10.1007/s40121-021-00455-1. Epub 2021 Jun 14. PMID 34125405
- [Derived] Mullhaupt B, Semela D, Ruckstuhl L, Magenta L, Clerc O, Torgler R, Negro F, Semmo N. Real-world effectiveness and safety of glecaprevir/pibrentasvir therapy in patients with chronic hepatitis C virus infection in Switzerland. Swiss Med Wkly. 2021 Jan 19;151:w20399. doi: 10.4414/smw.2021.20399. eCollection 2021 Jan 18. PMID 33516161
- See also: Related Info — http://rxabbvie.com